CLINICAL TRIAL: NCT07213583
Title: A Phase 2, Single Arm, Multicenter Study to Evaluate the Pharmacodynamics and Safety of Re-Treatment With ALXN2220 in Patients With Transthyretin Amyloid Cardiomyopathy
Brief Title: Study of Re-Treatment With ALXN2220 in Patients With ATTR-CM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Neurimmune AG (Industry)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NI006-102; 2025-520506-35-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-15; First posted 2025-10-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: Amyloid Transthyretin Cardiomyopathy
Keywords: Amyloid Depleter; ALXN2220; Transthyretin Amyloid Cardiomyopathy; Transthyretin amyloid (ATTR); Transthyretin (TTR); Amyloidosis; ATTR-CM
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALXN2220 (Experimental): Participants will receive ALXN2220 via intravenous (IV) infusion during the Active Treatment Period
  Interventions: Drug: ALXN2220

INTERVENTIONS:
Drug: ALXN2220 — Participants will receive ALXN2220 via IV infusion.

SUMMARY:
This is a Phase 2, single-arm, multicenter study to evaluate the pharmacodynamics and safety of re-treatment with ALXN2220 in previous participants of Study NI006-101.

DETAILED DESCRIPTION:
This is a Phase 2, single arm, multicenter study to evaluate the pharmacodynamics and safety of re-treatment with ALXN2220 in the patient population of previous participants in Study NI006-101.

The study will also explore changes in cardiac structure and function, and clinical function of this dosing regimen, as well as changes in cardiac amyloid load, structure and function during the treatment-pause since conclusion of Study NI006-101. The study consists of a Screening Period and a 48 week Active Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

* Must have received at least one dose of ALXN2220 in Study NI006-101

Exclusion Criteria:

* Suspected or known intolerance/allergy to proteins or any components of the study drug
* Treatment or study discontinuation in Study NI006-101 due to a treatment-related adverse event that was serious, severe or life-threatening (on Common terminology criteria for adverse events (CTCAE) scale)
* Any new or uncontrolled condition after completion of Study NI006-101 that could make the participant unsuitable for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 48 in ECV measured by cMRI | Baseline, Week 48
Change from Baseline to Week 48 in Heart Retention/Whole Body Retention measured by scintigraphy | Baseline, Week 48

SECONDARY OUTCOMES:
Incidence of TEAEs, including serious TEAEs | From Baseline up to Week 48
ALXN2220 serum concentrations | From Baseline up to Week 48
Incidence of Anti-Drug Antibodies | From Baseline up to Week 48

CONTACTS AND LOCATIONS:
Locations (6):
- France (3):
  - Hôpital Henri Mondor, Créteil
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - CHU Toulouse - Hôpital Rangueil, Toulouse
- Universitätsklinikum Heidelberg, Heidelberg, Germany
- University Medical Center Groningen, Groningen, Netherlands
- Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Spain

IPD SHARING:
Plan to Share IPD: Yes
Neurimmune has a public commitment to allow requests for study data and will be supplying protocol, results and plain language summaries.